CLINICAL TRIAL: NCT03287713
Title: Can Nasal High-Flow Oxygen Therapy Improve Oxygenation During Exercise, Optimizing Benefits of Pulmonary Rehabilitation in Patients With Interstitial Lung Disease (ILD) With Exercise Desaturation?
Brief Title: Can High-Flow Oxygen Therapy Improve Oxygenation During Exercise in ILD Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-OXI-2017-18
Record Dates: First submitted 2017-08-09; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Intersticial Lung Disease
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional oxygen (EPIDOC) (Active Comparator): Patients randomized in conventional oxygen (EPIDOC) group will perform a Pulmonary Rehabilitation Program. Oxygen will be titrated to flow needed to maintain SpO2 ≥ 90% during training with both systems.
  Interventions: Drug: oxygen therapy
- Nasal High-Flow oxygen therapy (EPIDOAF) (Active Comparator): Patients will be randomized in nasal High-Flow oxygen therapy (EPIDOAF) group will perform a Pulmonary Rehabilitation Program. Oxygen will be titrated to FiO2 needed to maintain SpO2 ≥ 90% during training with both systems.
  Interventions: Drug: oxygen therapy

INTERVENTIONS:
Drug: oxygen therapy — conventional nasal prongs vs nasal high flow oxygen during Pulmonary Rehabilitation in Interstitial Lung Disease.

SUMMARY:
Objectives: 1.- To compare the level of oxygenation achieved during muscular training with conventional oxygen systems (nasal cannulas) versus nasal High-flow oxygen therapy. 2.-To compare benefits achieved with both systems, in terms of: level of exercise during training; effort tolerance in the 6 minutes walking test (6MWT); improvement of dyspnoea and Health-related quality of life (HRQoL). And analyse the effects of nasal High-flow oxygen therapy on the acute exercise in a subgroup of patients.

Method: Multicentric randomized clinical trial. Patients with ILD in fibrotic phase who present oxygen desaturation during 6MWT (SpO2 mean ≤ 85%) will be included consecutively. Will be randomized in two groups: ILD patients with conventional oxygen (EPIDOC) and ILD patients with nasal High-Flow oxygen therapy (EPIDOAF). Both groups will perform a Pulmonary Rehabilitation Program. Oxygen will be titrated respectively to flow and FiO2 needed to maintain SpO2 ≥ 90% during training with both systems. Evaluation measures: SpO2 during training in both groups; dyspnoea (mMRC scale and CRQ dyspnoea); exercise capacity (6MWT) and HRQoL (self- administered KBILD questionnaire and SF36). In a subgroup of patients will be compared time of endurance exercise to evaluate the effects of nasal high-flow oxygen therapy in the acute exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age > 30 years old
* Diagnostic of ILD according to the national and international guidelines 23
* Being clinically stable the previous 4 weeks
* Acceptance to participate in the trial

Exclusion Criteria:

* Have been enrolled in a PR program in the last previous 6 months
* Respiratory Diseases other than ILD or severe comorbidities
* Osteoarticular diseases which don't allow training
* End-stage ILD, treatment with opiates or survival < 6 months
* Cognitive alterations that preclude colaboration

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Level of Sat O2 achived (in %) by conventional O2 vs nasal high flow oxygen during Pulmonary Rehabilitation | 8 weeks
  To compare the level of oxygenation (in SatO2 %) achieved by conventional oxygen therapy and nasal high flow oxygen therapy during muscular training program in patients with ILD measured by pulseoxymetry.

SECONDARY OUTCOMES:
Dyspnoea (benefits in borg scale) DURING effort. | 8 weeks
  To compare the benefits in dyspnoea achieved by both systems in terms of Effort level during the training period measured by Borg Scale.
Effort capacity (Benefits in terms of meters walked in the 6mwt). | 8 weeks
  To compare the benefits achieved by both systems in terms of Effort tolerance after PR program, evaluated with the 6 minut waking test (6WT), in meters.
Basal dyspnoea (mesured by mMRC scale). | 8 weeks
  To compare the benefits achieved by both systems in terms of Improvement in basal dyspnea measured by mMRC scale.
Basal dyspnoea (mesured by the dyspnoea area of CRQ questionnaire). | 8 weeks
  To compare the benefits achieved by both systems in terms of Improvement in basal dyspnea measured by the dyspnoea area of CRQ questionnaire.
Quality of life (SF36 questionnaire). | 8 weeks
  To compare the benefits achieved by both systems in terms of Improvement in HRQoL (with SF36 questionnarire).
Quality of life (KBILD questionnaire). | 8 weeks
  To compare the benefits achieved by both systems in terms of Improvement in HRQoL (with KBILD questionnaire).